CLINICAL TRIAL: NCT02596282
Title: A Randomized Trial of the Acceptability and Safety of Early Infant Male Circumcision (EIMC) Conducted by Nurse Midwives and Clinical Offices Using the Mogen Clamp
Brief Title: Enhanced Provision of Male Circumcision (MC) for HIV Prevention, Rakai, Uganda
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Rakai Health Sciences Program (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Principal Investigator, Ronald Gray, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00004524
Record Dates: First submitted 2015-10-23; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Neonatal Male Circumcision
Keywords: neonatal male circumcision; Clinical officers vs Nurse midwives; Rakai, Uganda; acceptability and safety of neonatal male circumcision

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical Officer (CO), (Active Comparator): COs were trained and provided neonatal male circumcision under topical anesthesia using the Mogen clamp
  Interventions: Procedure: Neonatal circumcision under topical anesthesia
- Nurse Midwife (NMW) (Experimental): NMWs were trained and provided neonatal male circumcision under topical anesthesia using the Mogen clamp
  Interventions: Procedure: Neonatal circumcision under topical anesthesia

INTERVENTIONS:
Procedure: Neonatal circumcision under topical anesthesia — The standard procedure for neonatal circumcision is as follows: combined analgesia was topical 2.5% lidocaine and 2.5% prilocaine <1 gm applied 60 minutes and 40mg acetaminophen suppository 30 minutes prior to surgery. Infants were given a 24% sucrose solution pacifier if needed. Infants under 2 weeks of age received subcutaneous Vitamin K 1 mg. The perineum cleaned, and the penis swabbed with povidone iodine. Hemostats were applied at 3 and 9 o'clock positions and the glans pushed down. Traction was applied before placing the Mogen clamp, the clamp was closed for 5 minutes and the foreskin removed with a scalpel.
  Petroleum jelly (e.g., Vaseline) was applied to the glans and the wound covered with sterile gauze. Infants were observed for one hour. Mothers were instructed in wound care.
  Other Names: Mogen clamp; Pre-operative analgesia

SUMMARY:
Background: Medical male circumcision (MMC) for HIV prevention is a priority in 14 East and Southern African countries, and the long-term sustainability of MMC programs could best be achieved by early infant male circumcision (EIMC.) However, the acceptability and safety of EIMC provided by non-physicians is unknown.

Methods: We conducted a trial of EIMC using the Mogen clamp provided by newly trained clinical officers (CO) and nurse midwives (NMWs) in 4 health centers in rural Rakai, Uganda. 501 healthy neonates aged 1-28 days with normal birth weight and gestational age were randomized to CO (n=256) and NMWs (n=245), and were followed up at 24 hours, 7 and 28 days. Combined analgesia was provided by paracetamol suppository, Eutectic Mixture of Local Anesthetics (EMLA) cream and a 24% sucrose solution.

DETAILED DESCRIPTION:
The objective was to assess the acceptability and safety of neonatal male circumcision performed by clinical officers (equivalent to US physician assistants) and nurse midwives, using the Mogen clamp.

This was a randomized, blinded trial of circumcision using the Mogen clamp under topical anesthesia in healthy male infants aged 1-28 days, with normal birth weight and gestational age, performed by trained clinical officers or nurse midwives, randomized 1:1 in Rakai District, Uganda.

Mothers of male infants born in 4 health centers were invited to participate and signed an informed consent for screening and enrollment. Infants were screened on enrollment prior to randomization (1;1) to clinical officer and nurse midwife circumcision providers.

Follow up was via a phone call at 24 hours, 7 days and 4 weeks post-circumcision.

ELIGIBILITY:
Inclusion Criteria:

* age 1-28 days
* birth weight >= 2,500 gm
* gestational age >=37 weeks
* no illness. normal temperature
* no genital anatomic abnormality

Exclusion Criteria:

* age >28 days
* birth weight <2,500 gm
* gestational age <37 weeks
* Ill health
* genital abnormality

Ages: 1 Day to 28 Days | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 501 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Adverse events related to circumcision | 4 weeks
  Adverse events graded as mild, moderate and severe
Acceptability as measured by the proportion of mothers directly informed about the study who consented to enroll in the trial | through study completion, an of 1 year
  Proportion of registered mother-child pairs in which the male infant was circumcised
Wound healing | 4 weeks
  Completed wound healing (clean intact scar without a scab or stitch sinus)

SECONDARY OUTCOMES:
Procedure time | Less than 15 minutes
  Length of time from preoperative prep to completion
Parental satisfaction | 4 weeks
  Mother's report of satisfaction with the procedure
Neonatal pain scale (NIPS) | During surgery
  based of facial expression, crying, breathing patterns, movement of arms and legs, and state of arousal. NIPS scores 0 were classified as no pain, scores 1-2 mild, scores 3-4 as moderate and >4 as severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Gray, MD MSc, Principal Investigator — Johns Hopkins Bloomberg School of Public Health

REFERENCES:
- [Derived] Kankaka EN, Murungi T, Kigozi G, Makumbi F, Nabukalu D, Watya S, Kighoma N, Nampijja R, Kayiwa D, Nalugoda F, Serwadda D, Wawer M, Gray RH. Randomised trial of early infant circumcision performed by clinical officers and registered nurse midwives using the Mogen clamp in Rakai, Uganda. BJU Int. 2017 Jan;119(1):164-170. doi: 10.1111/bju.13589. Epub 2016 Sep 6. PMID 27597563